CLINICAL TRIAL: NCT00944437
Title: Noninvasive Ventilation For Postoperative Acute Respiratory Failure: Comparison of Conventional Helmet With a Novel Full-Face Mask.
Brief Title: Continuous Positive Airway Pressure (CPAP) Ventilation Using a Novel Full-Face Mask Versus Conventional Helmet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to reach expected enrollment by anticipated dates.
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Guido Fanelli, Professor of Anesthesiology and Director, Anesthesia, Critical Care and Pain Medicine, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICU-ICU-02
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Respiratory Insufficiency; Respiratory Distress Syndrome, Adult; Chronic Obstructive Pulmonary Disease; Pulmonary Edema
Keywords: Ventilation, Mechanical; Positive-Pressure Respiration; Continuous Positive Airway Pressure
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Pulmonary Disease, Chronic Obstructive; Pulmonary Edema; Respiratory Aspiration | interventions — Head Protective Devices; Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helmet (Active Comparator): Patients in this group will receive continuous positive airway pressure delivered through a helmet connected to a high-flow reservoir system.
  Interventions: Device: Helmet
- Mask (Experimental): Patients in this group will receive continuous positive-airway pressure delivered through a novel full-face mask connected to a high-flow system. Expiratory pressure will be maintained using an expiratory valve connected to a T-tube.
  Interventions: Device: Full-face mask

INTERVENTIONS:
Device: Helmet — Continuous positive airway pressure for up to 24 h. Initial pressure will be 5 cmH2O, and will be increased by 2-3 cmH2O up to 10 cmH2O, in order to maintain SpO2 ≥90%.
  Other Names: Continuous Positive Airway Pressure; Noninvasive Ventilation; 4-Vent helmet (Rüsch, Germany)
  Arms: Helmet
Device: Full-face mask — Continuous positive airway pressure for up to 24 h. Initial pressure will be 5 cmH2O, and will be increased by 2-3 cmH2O up to 10 cmH2O, in order to maintain SpO2 ≥90%.
  Other Names: Continuous Positive Airway Pressure; Noninvasive Ventilation; Novastar mask (Dräger GmbH, Lubeck, Germany)
  Arms: Mask

SUMMARY:
The aim of this study is to compare two methods of delivery of noninvasive mechanical ventilation (NIV).

Since patient compliance and mechanical characteristics of the delivery devices are two fundamental variables in the success of NIV during acute respiratory failure, our hypothesis is that an improved patient-ventilator interface may improve the efficacy of therapy.

DETAILED DESCRIPTION:
Noninvasive ventilation (NIV) is the delivery of ventilatory support without the need for an invasive artificial airway. The use of noninvasive positive-pressure ventilation (NPPV) in acute respiratory failure has been steadily increasing for intensive care unit (ICU) patients. Noninvasive ventilation can often eliminate the need for intubation or tracheostomy and preserve normal swallowing, speech, and cough mechanisms. Discomfort of the device is one of the reason for the failure of NIV (30-40% of the cases).

The Novastar oro-nasal mask (Dräger Medical, Lubeck, Germany) is a flexible, transparent mask shell with a fine silicone gel cushion which adapts to the wearer's face. The pliable ring embedded inside the flexible clear shell allows the mask to be bent and adjusted to fit the patient's face (customized fit), while minimizing leakages. The mask has magnetic, self aligning clips for capture and secure fastening of the mask headgear. The magnetic clips are self-aligning.

The transparent flexible helmet for NIV (Rüsch 4-Vent, Teleflex Medical Europe, Athlone, Ireland) is fixed with two straps passing through each armpit. The braces are protected by hydrocolloid strips to prevent axillary decubitus. It is important to chose the right size of the helmet to avoid air leakages in the neck region. Two filters in the in- and expiratory way are necessary to reduce noise.

Different devices may lead to varying degrees of discomfort and, thus, improve compliance. Better tolerability of NIV may improve its efficacy. Therefore, we planned this randomized controlled trial to investigate whether different modalities of NIV delivery may affect therapeutical efficacy.

No randomized trials have compared helmets to the NOVASTAR full-face masks. This randomized, controlled study aims to assess whether the new full face mask improves gas exchange in patients admitted to ICU because of acute postoperative respiratory failure.

METHODS

Patients meeting criteria for NIV cycles will be enrolled in this trial. Informed written consent requirements were waived by the Internal Review Board since enrollment criteria meet common clinical guidelines and the two devices are both widely available (and approved for this indication).

Enrollment criteria are:

* Ongoing or recent history of respiratory failure (either primary or secondary)
* PaO2 <60 mmHg if breathing room air or PaO2/FiO2 <300 mmHg if receiving supplemental oxygen
* Acute dyspnea with respiratory rate >25 bpm and accessory muscle recruitment and/or paradoxical abdominal breathing

Patients will be excluded if:

* Refusing NIV
* Comatose (Glasgow Coma Scale <8) or unable to maintain a patent airway
* Hemodynamically unstable (systolic blood pressure <80 mmHg on recruitment, or receiving vasopressors/inotropes; ongoing angina/myocardial infarction; newly-developed arrhythmia with hemodynamic impact)
* Having recently (≤2 weeks) undergone oesophageal or upper respiratory tract surgery

Upon enrolment, patients will be randomized to receive NIV via one of the two available interfaces. In group H (for "helmet"), the continuous positive pressure is obtained by a high influx of fresh gases (air + oxygen) flowing through a high-compliance reservoir, with a positive end-expiratory pressure valve limiting outflow. In the M ("oral-nasal mask") group the same flow scheme is obtained using a T-tube attached to the mask. Patients' heads will be elevated to about 45° in both groups.

In both groups continuous positive airway pressure (CPAP) will be instituted at 5 cmH2O. Pressure will be increased by increments of 2-3 cmH2O until a maximum of 10 cmH2O in order to reach a peripheral blood oxygen saturation (SpO2) ≥ 90% with the lowest FiO2 possible.

Noninvasive ventilation will be ideally maintained for up to 24 h. Patients will be asked to wear the helmet/mask as long as possible. During ventilation-free periods, which will be maintained as short as possible, patients will receive 50% oxygen supplementation. The criteria for success of therapy and discontinuation of NIV will be a reversal of all criteria listed above for enrollment.

Criteria for NIV failure and subsequent intubation and mechanical ventilation will be:

* Coma (Glasgow Coma Scale <8) or inability to maintain a patent airway
* Hemodynamic instability (systolic blood pressure <80 mmHg on recruitment, or receiving vasopressors/inotropes; ongoing angina/myocardial infarction; newly-developed arrhythmia with hemodynamic impact)
* Intolerance to the interface
* Patient's inability to mobilize secretions
* PaO2/FiO2 ratio <140 mmHg after ≥1 h of ventilation

MAIN ENDPOINT AND SAMPLE SIZE

Arterial blood gas analyses will be performed upon enrollment, after 1 h, and after 24 h from enrollment. The null hypothesis of the study is that there will be no difference in the mean PaO2/FiO2 values between the two groups at 24 h. We will consider as clinically and statistically significant a difference of ≥50±60 mmHg between the groups.

A total of 50 patients will be enrolled. Sample size calculations are based on the assumption of a 5% risk of type I error and a 20% risk of type II error, while accounting for a 10-15% attrition rate.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing or recent history of respiratory failure (either primary or secondary)
* PaO2 <60 mmHg if breathing room air or PaO2/FiO2 <300 mmHg if receiving supplemental oxygen
* Acute dyspnea with respiratory rate >25 bpm and accessory muscle recruitment and/or paradoxical abdominal breathing

Exclusion Criteria:

* Refusing noninvasive ventilation
* Comatose (Glasgow Coma Scale <8) or unable to maintain a patent airway
* Hemodynamically unstable (systolic blood pressure <80 mmHg on recruitment, or receiving vasopressors/inotropes; ongoing angina/myocardial infarction; newly-developed arrhythmia with hemodynamic impact)
* Having recently (≤2 weeks) undergone oesophageal or upper respiratory tract surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Differences in PaO2/FiO2 ratio with respect to baseline (before NIV) values. | 24 h

SECONDARY OUTCOMES:
PaO2/FiO2 improvement at 1 h after beginning of ventilation. | 1 h after enrollment
Arterial carbon dioxide partial pressure (PaCO2) | At 1 and 24 h post-enrollment
Arterial blood pressure and incidence of hypotension (systolic blood pressure <90 mmHg or mean arterial blood pressure <60 mmHg) | Up to 24 h post-enrollment
Need for intubation | Up to 24 h post-enrollment
Intensive care unit stay | Up to 30 days
In-hospital mortality | Up to 30 days
Device-related complications: pressure sores, skin necrosis, air leak, eye inflammation, gastric distension. | Up to 24 h post-enrollment
Patient's rating of comfort with the device. Numerical rating scale ranging from 1 (unbearable) to 5 (very good.) | At 1 and 24 h post-enrollment
Success rate of NIV as delivered with either helmet or full-face mask. Success is defined as ≥50 mmHg improvement of PaO2/FiO2 ratio. | 24 h from initiation of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Study Chair — Dept. of Anesthesiology and Critical Care Medicine, University of Parma, Italy; Maria Barbagallo, MD, Principal Investigator — UO II Anestesia, Rianimazione e Terapia Antalgica, Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- University and Hospital of Parma (Azienda Ospedaliero-Universitaria di Parma), Parma, PR, Italy

REFERENCES:
- [Background] Appendini L, Patessio A, Zanaboni S, Carone M, Gukov B, Donner CF, Rossi A. Physiologic effects of positive end-expiratory pressure and mask pressure support during exacerbations of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1994 May;149(5):1069-76. doi: 10.1164/ajrccm.149.5.8173743.
- [Background] Celikel T, Sungur M, Ceyhan B, Karakurt S. Comparison of noninvasive positive pressure ventilation with standard medical therapy in hypercapnic acute respiratory failure. Chest. 1998 Dec;114(6):1636-42. doi: 10.1378/chest.114.6.1636. PMID 9872200
- [Background] Chadda K, Clair B, Orlikowski D, Macadoux G, Raphael JC, Lofaso F. Pressure support versus assisted controlled noninvasive ventilation in neuromuscular disease. Neurocrit Care. 2004;1(4):429-34. doi: 10.1385/NCC:1:4:429. PMID 16174945
- [Background] Collaborative Research Group of Noninvasive Mechanical Ventilation for Chronic Obstructive Pulmonary Disease. Early use of non-invasive positive pressure ventilation for acute exacerbations of chronic obstructive pulmonary disease: a multicentre randomized controlled trial. Chin Med J (Engl). 2005 Dec 20;118(24):2034-40. PMID 16438899
- [Background] Keenan SP, Sinuff T, Cook DJ, Hill NS. Does noninvasive positive pressure ventilation improve outcome in acute hypoxemic respiratory failure? A systematic review. Crit Care Med. 2004 Dec;32(12):2516-23. doi: 10.1097/01.ccm.0000148011.51681.e2. PMID 15599160
- [Background] Kramer N, Meyer TJ, Meharg J, Cece RD, Hill NS. Randomized, prospective trial of noninvasive positive pressure ventilation in acute respiratory failure. Am J Respir Crit Care Med. 1995 Jun;151(6):1799-806. doi: 10.1164/ajrccm.151.6.7767523.
- [Background] Masip J, Roque M, Sanchez B, Fernandez R, Subirana M, Exposito JA. Noninvasive ventilation in acute cardiogenic pulmonary edema: systematic review and meta-analysis. JAMA. 2005 Dec 28;294(24):3124-30. doi: 10.1001/jama.294.24.3124. PMID 16380593
- [Background] Meduri GU, Turner RE, Abou-Shala N, Wunderink R, Tolley E. Noninvasive positive pressure ventilation via face mask. First-line intervention in patients with acute hypercapnic and hypoxemic respiratory failure. Chest. 1996 Jan;109(1):179-93. doi: 10.1378/chest.109.1.179. PMID 8549183
- [Background] Meduri GU, Fox RC, Abou-Shala N, Leeper KV, Wunderink RG. Noninvasive mechanical ventilation via face mask in patients with acute respiratory failure who refused endotracheal intubation. Crit Care Med. 1994 Oct;22(10):1584-90. PMID 7924369